CLINICAL TRIAL: NCT06894628
Title: Genomics and Efficacy of Post-prostatectomy Salvage Radiotherapy With 'Extreme' Hypofractionation
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS248/24/IRE
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to validate the Decipher® genomic test, in which patients with biochemical recurrence after radical prostatectomy are treated with salvage radiotherapy with extreme hypofractionation (5+ Gy/fraction).

Validating the Decipher® genomic classifier based on the expression of 22 RNA genes in the prospective study "esSBRT"

DETAILED DESCRIPTION:
The esSBRT study ("Early salvage stereotactic radiotherapy (esSBRT) for biochemical recurrence after radical prostatectomy: a phase II study", RS1705/22 - opinion of the Central Ethics Committee IRCCS Lazio, Section IFO - Fondazione Bietti of 4 August 2022; NCT05667636) is a prospective phase II study developed and currently active at the Institute's Radiotherapy Unit, in which patients with biochemical recurrence of the disease after RP are treated on the prostatic lodge, and possibly on the pelvic lymph node stations, with hypofractionated radiotherapy in 5 sessions (5 Gy/fx). The aim is to be able to have a genomic classifier, such as Decipher®, for the patients enrolled in this protocol in order to complete the predictive evaluation. Furthermore, the project plans to profile PCa samples using a 'Comprehensive' panel of about 500 genes that allows to identify a specific molecular profile in the respective risk classes (low, intermediate and high) stratified with Decipher®. This evaluation would allow to identify the mutational structure of prostate cancer in an early stage of the disease, in particular by identifying the molecular alterations of the genes involved in homologous recombination repair (HRR) such as BRCA1, BRCA2, ATM, CDK12, CHEK2, PALB2.

The hypothesis is that the Decipher® risk classes (low, intermediate and high) correspond to a different risk of biochemical disease progression (defined as an increase in total PSA of 0.2 ng/ml above the nadir) independently or in addition to conventional clinicopathological criteria.

ELIGIBILITY:
Inclusion Criteria:

* patients enrolled at IRE under the "esSBRT" protocol (meeting the criteria of the same);
* patients who express written informed consent personally or through their legal representative/witness/curator/guardian/support administrator (participation in the ancillary study and data processing)

Exclusion Criteria:

* all exclusion criteria adopted for the "esSBRT" study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with biochemical recurrence after radical prostatectomy are treated with salvage radiotherapy with extreme hypofractionation (5+ Gy/fraction).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-11-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
Biochemical disease progression | 36 months
  The hypothesis that the Decipher® risk classes (low, intermediate and high) correspond to a different risk of biochemical disease progression will be measured as an increase in total PSA -prostate specific antigen- of 0.2 ng/ml above the nadir, independently or in addition to conventional clinicopathological criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Sanguineti, Doctor, Principal Investigator — IRCCS National Cancer Institute
Locations (1):
- IRCSS Regina Elena, Roma, Italy